CLINICAL TRIAL: NCT06112821
Title: Arteriovenous Fistula Maturation in Hemodialysis Patients With or Without Positive Antiphospholipid Antibodies : A Prospective Observational Cohort Study.
Brief Title: Arteriovenous Fistula Maturation in Hemodialysis Patients With or Without Positive Antiphospholipid Antibodies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Tatiana Besse-Hammer, Head of clinical trial unit, Brugmann University Hospital
Other Study IDs: AVF Maturation-aPL
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Data Collection; Medical Records; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- APL negative: Patients without persistent antiphospholipid antibodies (aPL) positivity
  Interventions: Other: Data collection in medical records; Other: Blood sampling
- APL positive: Patients with persistent antiphospholipid antibodies (aPL) positivity
  Interventions: Other: Data collection in medical records; Other: Blood sampling

INTERVENTIONS:
Other: Data collection in medical records — Data collection in medical records
Other: Blood sampling — Blood plasma and serum collection for biobanking. Future laboratory analyses encompass the analysis of endothelial dysfunction markers and other markers implicated in APS.

SUMMARY:
Hemodialysis (HD) is one of the most often used modalities of blood epuration in ends-stage renal diseases (ESRD) and requires the creation of a patent vascular access such as an arteriovenous fistula (AVF). Native AVF is associated with lower morbidity and mortality compared to hemocatheters.

AVF need a maturation process before its use. This process usually requires less than 6 weeks and consists in a complex vascular remodeling process. Maturation can be considered as the process leading to a newly created AVF being usable for hemodialysis; it encompasses enlargement and thickening of the draining fistula vein, increasing the blood flow in the absence of thrombosis and bleeding. According to the Kidney Disease Outcomes Quality Initiative (KDOQI) guidelines, AVF is considered matured (and therefore usable for HD) if 6 weeks after AVF creation surgery: (a) its diameter is at least 6mm, (b) its depth less than 6mm, (c) flow rate is at least 600ml/min and (d) its length is at least 6cm in order to allow a two needles cannulation. Delayed AVF maturation is a major complication that affects more than half of the AVF. It can be defined as the delay or absence of maturation according to KDOQI guidelines. The pathophysiology of delay or absence of AVF maturation is complex and multifactorial. It mainly involves thrombosis, stenosis, endothelial dysfunction, and hypercoagulability states.

In order to promote AVF maturation, the 2019 ERA-EDTA Clinical practice guidelines on peri- and postoperative care of native AVF and grafts for HD in adults, propose some medical treatments.

Antiphospholipid syndrome (APS) is an autoimmune disease, characterized by a prothrombotic state affecting both arterial and venous vasculature. Classification criteria have been proposed in 2006. In HD patient, up to 37% of patients have persistent aPL positivity. aPL positivity has been associated with vascular access thrombosis in retrospective studies.

The investigators performed a retrospective analysis of 113 patients in the HD department of the Brugmann Hospital between 01/01/2019 and 01/08/2019. Unpublished data that are currently under evaluation for publication, showed that the prevalence of APS and antiphospholipid antibody positivity (aPL) without APS, was 18.5% and the prevalence of APS was 10.7%. Antiphospholipid antibody positivity was identified as a risk factor for delayed AVF maturation. In multivariate analysis, antiphospholipid antibody positivity and stenosis were both independent risk factors for delayed maturation. There is a statistically significant association between delayed native AVF maturation and antiphospholipid antibody positivity. This association was independent of arteriovenous stenosis. This data suggest a potential non-stenotic and/or non-thrombotic mechanism of aPL related delayed maturation of the AVF in HD patients. More interestingly, a significant association between aPL positivity (with or without antiphospholipid syndrome) and delayed AVF maturation was found. This association was independent of stenosis.

Considering this association between aPL and failure of native AVF maturation, the aim of the present study is to further evaluate this association in a prospective cohort and to further identify a potential treatment option in order to reduce the prevalence of this very common complication '(i.e. AVF delay or absence of maturation).

ELIGIBILITY:
Inclusion Criteria:

Incident patients with chronic kidney disease (CKD) on stage G3b to G5, not end-stage renal disease, according to KDIGO guidelines

Exclusion Criteria:

* Patient already on hemodialysis maintenance therapy, or switching from peritoneal dialysis to hemodialysis
* Arteriovenous fistula creation not feasible surgically or technically, or surgery contra-indicated
* Known thrombophilia other than antiphospholipid syndrome
* Active neoplasia
* aPL assays not relevant (treatment, inflammatory state, etc...)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident patients with chronic kidney disease (CKD) on stage G3b to G5, not end-stage renal disease, according to KDIGO guidelines and aged from 18 to 75 years old.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
AVF maturation status | 6 weeks
  AVF maturation status according to KDIGO guidelines, evaluated by means of ultrasound/doppler (outflow, diameter, stenosis and/or thrombosis)

SECONDARY OUTCOMES:
Functional primary patency of AVF | 1 year
  Time between of AVF first use and AVF complication necessitating intervention
Type of AVF complication AVF Thrombosis | 1 year
  Identification of AVF complication: thrombosis/stenosis/bleeding complications/intimal hyperplasia dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Brugmann University Hospital, Brussels, Belgium

REFERENCES:
- [Derived] Taghavi M, Jacobs L, Kaysi S, Dernier Y, Cubilier E, Chebli L, Laureys M, Collart F, Demulder A, Antoine MH, Nortier J. Assessment of Arteriovenous Fistula Maturation in Hemodialysis Patients with Persistently Positive Antiphospholipid Antibody: A Prospective Observational Cohort Study. Life (Basel). 2025 Jan 24;15(2):168. doi: 10.3390/life15020168. PMID 40003577